CLINICAL TRIAL: NCT06792760
Title: Interoception in Functional Movement Disorders: Clinical and Neurophysiological Predictors of the Effect of Physiotherapy
Brief Title: Additive Effects of Interoceptive Training to Physiotherapy in Functional Movement Disorders (interoPTfmd)
Acronym: interoPTfmd
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: General University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NW24-04-00456; 53/23 Grant AZV VES 2024 VFN (Other: Ethics Committee of the General University Hospital in Prague)
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Functional Neurological Disorder; Functional Movement Disorder
Keywords: Functional Movement Disorder; Interoception; Physiotherapy; Breathing techniques; Interoceptive training; Attention
MeSH Terms: conditions — Conversion Disorder | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Pragmatic, prospective, single-blind, interventional parallel arm clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FMD specific physiotherapy (Active Comparator): This arm will receive specific physiotherapy treatment for people with Functional Movement Disorder based on published recommendations.
  Interventions: Other: Physiotherapy
- FMD specific physiotherapy + specific breathing techniques (Experimental): This arm will receive specific physiotherapy treatment for people with Functional Movement Disorder based on published recommendations + specific breathing exercises as interoceptive training
  Interventions: Other: Physiotherapy; Other: Specific Breathing Techniques

INTERVENTIONS:
Other: Physiotherapy — The intervention will consist of 10 individual physiotherapy sessions delivered by a single physiotherapist trained in FMD. The physiotherapy programme will include education, movement retraining and a self-management plan.
Other: Specific Breathing Techniques — The intervention will include education and training in specific breathing techniques, which will be exercised by the patient as a self-management plan for over 5-10 minutes daily.
  Arms: FMD specific physiotherapy + specific breathing techniques

SUMMARY:
Functional movement disorder (FMD) is a common source of neurological disability that imposes a significant financial burden on healthcare systems. However, the heterogeneous manifestations of FMD and numerous associated non-motor symptoms, often fluctuating over time, present a challenge for developing effective treatment pathways. Although increasing evidence supports the efficacy of physiotherapy for FMD, the lack of predictors of treatment outcomes remains a significant obstacle to effectively managing FMD. The main hypothesis of this project is that abnormalities in interoceptive processing are responsible for variability in motor and non-motor symptoms and response to physiotherapy. Interoception describes the afferent signalling, central processing, and mental representation of internal bodily signals. We hypothesize that worse performance on interoceptive tests will be associated with greater severity of motor and non-motor symptoms and worse quality of life. We also expect that patients with worse interoceptive performance and associated non-motor symptoms such as pain will particularly benefit from treatment techniques modulating interoception, such as specific breathing techniques. Therefore, to test our hypotheses, in this project, we will study interoceptive and attentional abnormalities of FMD and identify predictors of the effect of physiotherapy and interoceptive respiratory training.

DETAILED DESCRIPTION:
Functional Neurological Disorder (FND) is a poorly understood and prevalent disorder, making up 16% of outpatient neurology referrals. Patients with functional movement disorder (FMD), which is one of the most common subtypes of FND, are difficult to treat. While growing evidence highlights the effectiveness of physiotherapy for FMD, the absence of reliable predictors for treatment outcomes remains a major challenge in managing the condition effectively.

Our goal is to evaluate the interoceptive profile of individuals with FMD and establish a connection between interoceptive and attentional abnormalities, the type and severity of symptoms, and the response to treatment. The study will utilize the objective clinical and subjective evaluation of symptom severity along with behavioural, neurophysiological, and neuroimaging methods to provide a comprehensive set of measures of interoception and attention. fMRI will further elucidate the neural correlates of interoception and attention. These measures will be analyzed in a cohort of FMD patients and healthy controls to examine the relationship between interoception, attention, and the type, severity, and impact of motor and non-motor symptoms on quality of life.

Interoceptive and attentional measures will also be tested as markers of therapy outcomes in a prospective randomized controlled trial. Eighty FMD patients will be recruited to undergo FMD-specific physiotherapy, with one group receiving additional interoception training via a specific breathing technique (SBTs) protocol. Participants will be randomized to physiotherapy alone or physiotherapy plus SBTs, with clinical outcomes, interoceptive, and attentional measures assessed before and after treatment. This design will evaluate the interventions' impact and identify treatment outcome predictors.

Specific Aims Aim 1: To explore interoceptive mechanisms in FMD and their relationship to symptoms and treatment response.

1.1 Characterize interoceptive profiles (respiroceptive and cardioceptive sensitivity and metacognition) in FMD compared to healthy controls.

1.2 Investigate associations between interoception, motor symptoms, and pain. 1.3 Evaluate interoceptive sensitivity as a predictor of PT outcomes and the impact of SBTs on interoception and pain reduction.

1.4 Examine changes in interoceptive network activation (e.g., salience network) following PT, with or without SBTs.

Aim 2: To study attentional mechanisms in FMD and identify predictors of PT outcomes.

2.1 Assess distractibility as a predictor of PT outcomes. 2.2 Evaluate attentional measures during cognitive, emotional and oculomotor tasks and their relationship to FMD symptoms and PT outcomes.

2.3 Investigate changes in brain activation related to attentional processing and symptom control.

Aim 3: To evaluate the additive effects of specific breathing techniques (SBTs) on physiotherapy outcomes in FMD.

3.1 Compare outcomes between patients receiving PT alone and PT plus SBTs. 3.2 Assess whether SBTs enhance interoception and improve symptoms and HRQoL.

Methods:

Aim 1. Interoceptive sensitivity, metacognition, and attention will be evaluated using psychophysical tasks, fMRI, and eye-tracking to explore their relationship with symptoms and treatment outcomes in FMD.

Aim 2: Attentional mechanisms, including distractibility, will be assessed through clinical tasks, neurophysiological recordings, and fMRI to identify predictors of physiotherapy outcomes.

Aim 3: The effects of SBTs as an adjunct to physiotherapy will be evaluated using clinical scales for motor and non-motor symptoms, alongside quality-of-life and psychological measures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* clinically established diagnosis of Functional Movement Disorder according to Gupta and Lang criteria

Exclusion Criteria:

* age <18 years
* inability to complete questionnaires because of language difficulties
* severe learning disabilities or cognitive impairment
* major psychiatric or organic neurological comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impressions (CGI) scale - patient rated | pre-treatment (baseline), one week after the last intervention, 6-month follow-up, 12-month follow-up
  Clinical Global Impressions (CGI-I) scale, patient-rated, is a 5-point scale evaluating improvement from 'very much improved' to 'very much worse'. 'Very much improved' indicates a better outcome.

SECONDARY OUTCOMES:
Clinical Global Impressions (CGI) - clinician rated scale | one week after the last intervention, 6-month follow-up, 12-month follow-up
  Adapted Patient Clinical Global Impression Improvement (CGI-I) scale rated by the outcome assessor is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
36-item Short Form Survey (SF-36) | pre-treatment (baseline), one week after the last intervention, 6-month follow-up, 12-month follow-up
  The 36-item Short Form Health Survey (SF-36) is a self-report test assessing functional ability. Scores range from 0 to 100, with higher scores indicating better outcomes.
Fibromyalgia Survey Questionnaire | pre-treatment (baseline), one week after the last intervention, 6-month follow-up, 12-month follow-up
  The Widespread Pain Index (WPI) and Somatic Symptom (SS) score are evaluated using the Fibromyalgia Survey Questionnaire. The WPI score ranges from 0 to 19 and assesses the distribution of pain across the body, while SS scores evaluate the intensity of associated symptoms. Higher scores indicate a worse outcome.
The Simplified Functional Movement Disorders Rating Scale (S-FMDRS) | pre-treatment (baseline), one week after the last intervention, 6-month follow-up, 12-month follow-up
  The Simplified Functional Movement Disorders Rating Scale (S-FMDRS), a clinician-rated scale, assesses the severity of motor disorder symptoms across seven body regions. Scores range from 0 to 54, with higher scores indicating greater severity.

OTHER OUTCOMES:
Work and Social Adjusment Scale (WSAS) | pre-treatment (baseline), 6-month follow-up, 12-month follow-up
  The Work and Social Adjustment Scale (WSAS) is used to assess participants' socioeconomic conditions. Each item is rated on a 9-point scale from 0 (no impairment at all) to 8 (very severe impairment), with the total score ranging from 0 to 40. Lower scores indicate a better outcome.
Illness belief and understanding and confidence in the diagnosis | pre-treatment (baseline)
  A patient-rated measure will assess illness belief and understanding using a 5-point Likert scale and confidence in their diagnosis using a 3-point Likert scale. These measures will be evaluated as a potential predictor of physiotherapy outcomes in patients with FMD.
Readiness for treatment | pre-treatment (baseline)
  Readiness for treatment will be assessed by patients using a 5-point Likert scale and evaluated as a potential predictor of therapy outcomes.
Distractibility assessment of motor symptoms | pre-treatment (baseline) and one week after the last intervention
  The effects of competitive motor or cognitive tasks on abnormal movements (2 = complete suppression, 1 = variable/incomplete suppression, 0 = non-distractible) and performance quality in the competitive task (2 = good, 1 = effortful/impaired, 0 = unable) will be recorded. This measure will be evaluated as a potential predictor of physiotherapy outcomes in FMD.
Adapted Patient Health Questionnaire-15 (PHQ-15) | pre-treatment (baseline), one week after the last intervention, 6-month follow-up, 12-month follow-up
  Adapted Patient Health Questionnaire 15 (PHQ15) will be used as a measure of somatic symptom (physical) severity. Relationship between changes in subjectively reported symptom sevrity subscores, interoceptive measures and fMRI data pre and post treatment will be analysed.
Fatigue Severity Scale (FSS) | pre-treatment (baseline), one week after the last intervention, 6-month follow-up, 12-month follow-up
  The Fatigue Severity Scale (FSS) is a 9-item self-report test that assesses the functional impact and severity of physical and mental fatigue experienced over the past week. Each item is scored on a scale from 1 to 7, and the total score is calculated as the average of the item scores. Higher scores indicate a worse outcome. Relationship between changes in FSS scores, interoceptive measures and fMRI data pre and post treatment will be analysed.
Multidimensional Inventory of Subjective Cognitive Impairment (MISCI) | pre-treatment (baseline), one week after the last intervention, 6-month follow-up, 12-month follow-up
  The Subjective Cognitive Impairment Scale (MISCI) will be used to evaluate participants' cognitive functioning. It consists of 10 items, with scores ranging from 10 to 50. Higher scores indicate a worse outcome. Relationship between changes in MISCI scores, interoceptive measures and fMRI data pre and post treatment will be analysed.
Beck Depression Inventory (BDI-II) | pre-treatment (baseline), one week after the last intervention, 6-month follow-up, 12-month follow-up
  Beck Depression Inventory (BDI-II), 21-item scale, assessing depressive symptoms over the last 14 days. Scores range from 20 to 80, with lower scores indicating a better outcome. Relationship between changes in BDI scores, interoceptive measures and fMRI data pre and post treatment will be analysed.
Generalized Anxiety Disorder 7-item (GAD-7) | pre-treatment (baseline), one week after the last intervention, 6-month follow-up, 12-month follow-up
  Generalised Anxiety Disorder 7 (GAD-7) will be used for evaluating participants' psychological conditions; scores from 0 to 21, higher scores mean a worse outcome. Relationship between changes in GAD-7 scores, interoceptive measures and fMRI data pre and post treatment will be analysed.
Trail Making Test (TMT) | pre-treatment (baseline)
  The Trail Making Test (TMT) - a computer-based eye-tracking test and a pen and paper version will measure attention, processing speed, and cognitive flexibility. In TMT-A, participants connect numbered circles sequentially, while in TMT-B, they alternate between numbers and letters. Completion time indicates cognitive performance, with longer times suggesting impairments. This measure will be evaluated as a potential predictor of physiotherapy outcomes in patients with functional movement disorders.
Multiscale Dissociation Inventory (MDI) | pre-treatment (baseline)
  The MDI is a 30-item self-report test of dissociative symptomatology with scores ranging 0 to 120. It measures six different types of dissociative responses (Disengagement, Identity Dissociation, Emotional Constriction, Memory Disturbance, and Depersonalization/Derealization). Higher scores indicate a worse outcome. It will be assessed as a potential predictor of therapy outcomes.
Maltreatment and Abuse Chronology of Exposure (MACE) | pre-treatment (baseline)
  The Maltreatment and Abuse Chronology of Exposure (MACE) is a self-report instrument designed to assess the severity and timing of exposure to ten types of maltreatment during childhood, with scores reflecting the degree of exposure. Higher scores indicate a greater severity and multiplicity of maltreatment experienced. It will be assessed as a potential predictor of therapy outcomes.
The Attention-Emotion task | pre-treatment (baseline), one week after the last intervention
  The Attention-Emotion Task is a video-based eye-tracking assessment (The Free Viewing Task) designed to evaluate saccadic, pupillary, and blink responses. Parameters tracked include baseline pupil size and changes in diameter, pupil constriction and dilation latencies, constriction and dilation velocities, saccadic eye movements, and blink responses. These measures provide quantitative insights into attention and emotional processing, which will provide insights into neural mechanisms underlying FMD.
Bayesian psychophysical interoceptive task | pre-treatment (baseline), one week after the last intervention
  A fully computer-controlled adaptive psychophysical estimation of respiroceptive and cardioceptive thresholds (success in correctly identifying respiratory resistance or delay in heartbeat feedback), as well as improved estimation of other signal-theoretic parameters such as sensitivity, bias, and metacognition which will provide insights into neural mechanisms underlying FMD.
fMRI - Interoceptive Awareness Task. | pre-treatment (baseline), one week after the last intervention
  A fMRI paradigm for characterizing the neural dynamics of interoceptive attention vs. a closely balanced exteroception task. Participants are required to judge whether the presented breath curve was delayed relative to the breath rhythm they perceived from their body. In the exteroceptive condition, participants are instructed to detect whether a dot flashed on the respiratory curve at any time when the breath curve was displayed. Changes in BOLD signal between the conditions will be compared. Pre- and post-treatment evaluation will be used to assess mechanisms underlying FMD.
fMRI - Distraction Task | pre-treatment (baseline), one week after the last intervention
  A fMRI distraction task developed in our lab estimates neural activity during attentional engagement in external stimuli relative to body focus (baseline condition). In the task, there are dynamic stimuli participants are requested to follow, the difficulty of the task is adjusted by varying the speed of the stimuli moving on the screen. The difficulty will be set individually on two levels (30% and 70% hit-rate) in a staircase procedure before fMRI to mitigate task difficulty effects. BOLD changes between conditions will be assessed. The pre and post-treatment assessment will provide insights into mechanisms underlying FMD.

CONTACTS AND LOCATIONS:
Overall Officials: Tereza Serranová, MD, PhD, Study Director — General University Hospital in Prague, Neurology department, Prague, Czech Republic, 12800
Locations (1):
- General University Hospital in Prague, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: "Beginning 1 year after publication with no end date"
Access Criteria: Anonymized data will be shared with other researchers based on reasonable request.